CLINICAL TRIAL: NCT07117916
Title: STRONGER 60+: Assessing the Clinical Effectiveness and Delivery of an Adapted FINGER Model for Brain Health in Primary Care
Acronym: STRONGER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Stiftelsen Stockholms Sjukhem (Other)
Responsible Party: Principal Investigator, Miia Kivipelto, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-01125
Record Dates: First submitted 2025-08-11; First posted 2025-08-12 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-08

CONDITIONS: Older Adults at High Risk for MCI; Older Adults With Mild to Moderate Level of Dementia
Keywords: Dementia prevention; Primary care; Clinical effectiveness; Randomized controlled trial
MeSH Terms: interventions — Exercise; Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised multidomain intervention (Experimental): The supervised intervention includes nutritional guidance, physical exercise, cognitive training, social engagement, and management of vascular and metabolic risk factors.
  Interventions: Behavioral: Supervised nutritional guidance, physical exercise, cognitive training, social engagement, and management of vascular and metabolic risk factors.
- Self-guided intervention (Active Comparator): Self-guided version of the intervention.
  Interventions: Behavioral: Supervised nutritional guidance, physical exercise, cognitive training, social engagement, and management of vascular and metabolic risk factors.

INTERVENTIONS:
Behavioral: Supervised nutritional guidance, physical exercise, cognitive training, social engagement, and management of vascular and metabolic risk factors. — In addition to health advice, participants in the intervention group will receive a structured, multidomain lifestyle program comprising nutritional guidance, physical exercise, cognitive training and social engagement, and monitoring and management of vascular and metabolic risk factors. The STRONGER 60+ intervention is based on the FINGER protocol and has been specifically adapted for primary care to enhance feasibility and scalability. Key adaptations include 1) delivering physical exercise sessions at external gym facilities rather than at primary care centers, and 2) shortening the intervention duration from two years to six months.

SUMMARY:
Background: The Finnish Geriatric Intervention Study to Prevent Cognitive Impairment and Disability (FINGER) was the first to show that multidomain lifestyle interventions can enhance brain health and reduce cognitive decline. However, the clinical effectiveness and delivery of the FINGER model within primary care settings remain unexplored. The aim of the STRONGER 60+ trial is to evaluate both the clinical effectiveness and real-world delivery of an adapted FINGER-based intervention in primary care.

Methods and analysis: This 6-month randomized controlled clinical effectiveness trial will be conducted in primary care and will include adults aged 60 and older with vascular or lifestyle-related risk factors for dementia. A total of 96 participants will be randomized to either a structured, supervised multidomain lifestyle intervention or a self-guided version of the same program. The intervention includes nutritional guidance, physical exercise, cognitive training, social engagement, and management of vascular and metabolic risk factors. Data will be collected at baseline, 6 months (primary endpoint), and 12 months post-randomization. The primary outcome is the change in a composite healthy lifestyle score at 6 months. In addition, the study will explore delivery processes and stakeholder (participant and healthcare professional) perspectives using both qualitative and quantitative methods.

ELIGIBILITY:
Inclusion Criteria:

Individuals aged 60 and older who express interest in the study will be pre-screened by the research team using the CAIDE (Cardiovascular Risk Factors, Aging, and Dementia) Risk Score. Those scoring ≥6-indicating elevated dementia risk-will be invited for an in-person screening visit to confirm eligibility. The CAIDE score (range: 4-15) is based on age, sex, education, systolic blood pressure, BMI, total cholesterol, and physical activity. Additional inclusion criteria are a Mini-Mental State Examination (MMSE) score of ≥24, and ability to walk independently indoors and outdoors (with or without a mobility aid).

Exclusion Criteria:

Exclusion criteria include diagnosed dementia and residence in a nursing home.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2026-08-01 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Composite healthy lifestyle score | Assessments are conducted at baseline, 6 months (primary endpoint), and 12 months post-randomization
  The primary outcome is a composite healthy lifestyle score based on four domains measured individually: dietary intake (Mediterranean Diet Adherence Screener ), physical activity (ActiGraph), cognitive and social engagement (combined self-reported), and cardiovascular risk burden (BMI, lipids, glucose, waist-to-hip ratio, and smoking status).

SECONDARY OUTCOMES:
Functioning and symptoms | Baseline, 6- and 12 months post randomization
  Physical function by Short Physical Performance battery (SPPB) and 10 meter walking test, Cognitive function by Mini Mental State Examination (MMSE), Geriatric Depression Scale (GDS15), Health Related Quality of Life (RAND-36), Pittsburg Sleep Quality Index (PSQI)

CONTACTS AND LOCATIONS:
Overall Officials: Miia Kivipelto, PhD, Professor, Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: No
The data to be collected will be available upon request. Requests for access can be directed to the Research Data Office (rdo@ki.se) at Karolinska Institutet, where they will be processed in accordance with relevant legislation. Access will require a data processing agreement or equivalent with the data recipient. This procedure complies with the General Data Protection Regulation, reflecting the high sensitivity of the data and the potential harm to individuals if made publicly available.